CLINICAL TRIAL: NCT00930618
Title: NOCETER, a Multicenter Double Blind Placebo-controlled Randomized Trial: Reduction of CEsareans in Post TERm Pregnancies: Impact of Outpatient Cervical Ripening With NO Donors
Brief Title: Reduction of Cesareans by Nitric Oxide (NO) Donors in Post Term Pregnancies
Acronym: NOCETER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P071212
Record Dates: First submitted 2009-06-29; First posted 2009-06-30 (Estimated); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Prolonged Pregnancy; Nulliparity
Keywords: Prolonged pregnancy; Nulliparity; Cervical ripening; Induced labor; Cesarean section
MeSH Terms: conditions — Pregnancy, Prolonged

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IMN (Experimental): Isosorbide mononitrate
  Interventions: Drug: IMN
- Placebo (Placebo Comparator): Administration of placebo of IMN
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IMN — Administration of 2 x 20 mg of isosorbide mononitrate at each administration with a maximum of three administrations
  Arms: IMN
Drug: Placebo — Administration of 2 X 20 mg of placebo of IMN at each administration with a maximum of three administration
  Arms: Placebo

SUMMARY:
The purpose of this trial is to determine whether cervical ripening with isosorbide mononitrate reduce caesarean section in women with post term pregnancies.

DETAILED DESCRIPTION:
The purpose of this trial is to determine whether cervical ripening with 40 mg of isosorbide mononitrate given intravaginally at 41+0, 41+2 and 41+4 weeks reduce cesarean section in nullipara with post term pregnancies. Treatments will be administered by midwifes in the maternity wards, women will be allowed to go back home in case of Bishop score<6. Otherwise labor will be induced with oxytocin. If undelivered at 41+5, women with Bishop score<6 will be induced with prostaglandins according to local protocols.

ELIGIBILITY:
Inclusion criteria :

* Age > or = 18 years old
* TAS > or = 95 mmHg
* Singleton
* Nulliparity
* Term > or = 41 weeks + 0 day
* Bishop score < or = 5
* Vertex presentation
* Intact membranes
* No contra-indications of the study treatment
* No maternal or fetal diseases which could indicate immediate labor induction
* Written informed consent

Exclusion criteria :

* Multiple pregnancy
* Multiparity
* Term < 41 weeks
* Bishop score > 5
* Breech presentation
* Rupture of the membranes
* Previous cesarean
* Indication to immediate labor induction
* Contraindications to isosorbide mononitrate
* No co-administration of antihypertensive drugs
* No social security

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1409 (Actual)
Dates: Start 2009-06; Primary Completion 2013-12 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Number of cesarean sections | 10 days

SECONDARY OUTCOMES:
Number of labor inductions | 10 days
Number of spontaneous labors | 10 days
Cesarean for failed labor induction | 10 days
Cesarean for FHR abnormalities | 10 days
Cesarean for arrested labor | 10 days
Mean time between randomisation and spontaneous labor | 10 days
Isosorbide mononitrate adverse effects | 10 days
Maternal satisfaction | 10 days
Neonatal morbidity | 10 days
Mean time between randomisation and delivery | 10 days
Mean duration of labor | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: François Goffinet, MD, PhD, Study Director — Scientific Responsible
Locations (1):
- Robert Debré Hospital, Paris, France

REFERENCES:
- [Result] Schmitz T, Fuchs F, Closset E, Rozenberg P, Winer N, Perrotin F, Verspyck E, Azria E, Carbonne B, Lepercq J, Maillard F, Goffinet F; Groupe de Recherche en Obstetrique et Gynecologie (GROG). Outpatient cervical ripening by nitric oxide donors for prolonged pregnancy: a randomized controlled trial. Obstet Gynecol. 2014 Dec;124(6):1089-1097. doi: 10.1097/AOG.0000000000000544. PMID 25415159